CLINICAL TRIAL: NCT03989544
Title: An Open Label, Randomized, Parallel Group Study to Evaluate the Pharmacokinetics of Tezepelumab Administered Subcutaneously Via Accessorized Pre Filled Syringe (APFS) or Autoinjector (AI) Compared With Vial and Syringe in Healthy Adult Subjects (PATH-BRIDGE)
Brief Title: A Study to Evaluate the Pharmacokinetics of Tezepelumab After Being Delivered by an Accessorized Pre Filled Syringe or Autoinjector Compared With Vial and Syringe in Healthy Adult Subjects
Acronym: PATH-BRIDGE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00012
Record Dates: First submitted 2019-06-16; First posted 2019-06-18 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: Pharmacokinetics; Human monoclonal antibody; Tezepelumab; Accessorized Pre-filled Syringe; Autoinjector
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Tezepelumab via Vial-and-syringe (Experimental): Participants will be randomized to a single dose of tezepelumab via SC administration with Vial-and-syringe
  Interventions: Biological: Tezepelumab
- Tezepelumab via APFS (Experimental): Participants will be randomized to a single dose of tezepelumab via SC administration with APFS
  Interventions: Biological: Tezepelumab
- Tezepelumab via AI (Experimental): Participants will be randomized to a single dose of tezepelumab via SC administration with AI
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection

SUMMARY:
This is a study to compare PK of tezepelumab exposure in healthy subjects by using vial and syringe, APFS, and AI.

DETAILED DESCRIPTION:
This study will be a single center, randomized, open label, parallel group study designed to compare tezepelumab PK exposure in healthy subjects following single subcutaneous (SC) administration of a fixed dose of tezepelumab by using vial and syringe, APFS, or AI. A total of 315 subjects will be randomized to receive a single, fixed dose of tezepelumab administered SC using vial-and-syringe, APFS, or AI at 1 of 3 injection sites: abdomen, thigh or upper arm. Separate randomization lists will be produced for each weight group (50 to < 70 kg, 70 to < 80 kg, 80 to 90 kg), and within each of the 3 weight groups, subjects will be randomized 1:1:1:1:1:1:1:1:1 to 1 of the 9 combinations of treatment (vial-and-syringe, APFS, or AI) with injection site (abdomen, thigh, upper arm). Within each weight group, at least 36 subjects will be randomized resulting in at least 12 subjects per treatment group (device) within each weight group.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 65 years (inclusive) at the Screening Visit, with suitable veins for repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit (Day 1) and must not be lactating.
4. Females of childbearing potential who are sexually active must use a highly effective method of contraception from the Screening Visit and must agree to continue using such precautions for 16 weeks after the dose of Investigational Medicinal Product (IMP). Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.
5. Have a body mass index between 18.5 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 90 kg inclusive.
6. Intact normal skin without potentially obscuring tattoos, scars, pigmentation or lesions on the skin area intended for injection (abdomen, thigh, upper arm).

Exclusion Criteria:

1. History of any clinically significant disease or disorder.
2. History of anaphylactic reaction to biologic therapy.
3. Acute upper or lower respiratory infection requiring antibiotics or antiviral medications.
4. History of tuberculosis.
5. History of known immunodeficiency disorder, including a positive human immunodeficiency virus, or the subject is taking antiretroviral medications.
6. Receipt of any marketed or investigational biologic agent within 4 months or 5 half lives prior to the Screening Visit.
7. Current smokers or those who have smoked or used nicotine products including e-cigarettes within the 3 months prior to the Screening Visit.
8. History of cancer:

   Subjects who have had basal cell carcinoma or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to the Screening Visit.

   Subjects who have had other malignancies including breast cancer are eligible provided that curative therapy was completed at least 5 years prior to the Screening Visit.
9. Subjects who have previously received tezepelumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The area under the time concentration curves from zero to infinity (AUCinf) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To compare the AUCinf following single SC administration of tezepelumab using Vial-and-syringe, APFS, and AI.
The maximum observed concentration (Cmax) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To compare the Cmax following single SC administration of tezepelumab using vial-and-syringe, APFS, and AI.

SECONDARY OUTCOMES:
The areas under the time concentration curves from zero to last observation (AUClast) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To determine the AUClast following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.
Time to Cmax (tmax) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To determine time to Cmax (tmax) following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.
Terminal phase elimination half life (t½λz) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To determine t½λz following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.
Apparent systemic clearance (CL/F) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To determine CL/F following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.
Apparent terminal phase volume of distribution (Vz/F) | At Days 1, 2, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  To determine Vz/F estimated by non compartmental analysis following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.
Presence of ADAs to tezepelumab | At Day 1, 15, 29, 71 and 113
  To evaluate the immunogenicity of single dose tezepelumab administered SC using Vial-and-syringe, APFS and AI
Number of subjects with adverse events (AEs)/ serious adverse events (SAEs) | From screening (Day -28) to follow up period (Day 113)
  To determine the number of subjects with AEs/SAEs following single dose SC administration of tezepelumab using vial and syringe, APFS and AI.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Derived] Corren J, Ambrose CS, Salapa K, Roseti SL, Griffiths JM, Parnes JR, Colice G. Efficacy of Tezepelumab in Patients with Severe, Uncontrolled Asthma and Perennial Allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4334-4342.e6. doi: 10.1016/j.jaip.2021.07.045. Epub 2021 Aug 3. PMID 34358701
- [Derived] Zheng Y, Abuqayyas L, Megally A, Fuhr R, Salapa K, Downie J, Colice G. Tezepelumab Pharmacokinetics, Safety, and Tolerability After Administration via Vial-and-syringe, Accessorized Prefilled Syringe, or Autoinjector: A Randomized Trial in Healthy Volunteers. Clin Ther. 2021 Jan;43(1):142-155.e5. doi: 10.1016/j.clinthera.2020.11.014. Epub 2020 Dec 27. PMID 33380362